CLINICAL TRIAL: NCT00183560
Title: Prevention of Relapse in Recurrent Depression With MBCT
Brief Title: Preventing Depression Relapse With Mindfulness-Based Cognitive Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Zindel Segal, Psychologist / Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R01MH066992 (NIH); R01MH066992 (NIH); DSIR 83-ATP
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Depression
Keywords: Depression Recurrence; Drug Therapy; Cognitive Therapy; Relapse; Antidepressants
MeSH Terms: conditions — Depression; Recurrence | interventions — Mindfulness-Based Cognitive Therapy; Antidepressive Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Participants will receive mindfulness based cognitive therapy
  Interventions: Behavioral: Mindfulness based cognitive therapy (MBCT)
- 2 (Active Comparator): Participants will receive maintenance antidepressant pharmacotherapy
  Interventions: Drug: Antidepressants
- 3 (Placebo Comparator): Participants will receive placebo plus clinical management
  Interventions: Drug: Placebo plus clinical management

INTERVENTIONS:
Behavioral: Mindfulness based cognitive therapy (MBCT) — Following antidepressant discontinuation, participants receive MBCT, an 8-week group program that integrates aspects of cognitive therapy and mindfulness meditation.
  Other Names: MBCT
  Arms: 1
Drug: Antidepressants — Participants continue on dosage of the antidepressant that was used to achieve clinical remission.
  Other Names: Antidepressant medication
  Arms: 2
Drug: Placebo plus clinical management — Following discontinuation of active antidepressant, participants are placed onto the placebo and clinical management regimen.
  Other Names: Placebo and Clinical Management
  Arms: 3

SUMMARY:
This study will determine the effectiveness of mindfulness-based cognitive therapy (MBCT) in preventing depression relapse.

DETAILED DESCRIPTION:
Depression is a serious condition that can cause significant social and emotional problems and reduce the overall quality of life. Relapses in depressive episodes are common and may result in a patient's reluctance to follow a treatment regimen, thus making the episode more severe. Safe and effective therapies to prevent depression relapse are needed. This study will compare three different approaches to determine which is most effective in preventing relapses in depressive episodes.

This study will comprise 2 parts. In Part 1, all participants will receive antidepressant medication for 6 months. Participants whose depression symptoms do not improve will complete their study participation at the end of Part 1. Participants who respond to their regimen will be enrolled in Part 2. This part will last 18 months. During Part 2, participants will be randomly assigned to one of three groups. Participants in Group 1 will continue the drug regimen they began in Part 1. Participants in Group 2 will discontinue their antidepressants and attend an 8-week relapse prevention program. This MBCT program is designed to help participants learn skills that can increase their awareness and change their reaction to stressful events. Participants in Group 3 will have their antidepressant medication from Phase 1 switched to a placebo without their knowledge. Self-report scales will be used to assess the depressive symptoms of participants at the beginning of the study, at the end of Phase 1, and at the end of the study, after Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM criteria for recurrent major depressive disorder, defined as at least one major depressive episode within 3 years prior to study entry AND at least 2 months of normal functioning following the episode

Exclusion Criteria:

* Depression secondary to a concurrent medical disorder
* Current use of medication that could cause depressive symptoms
* A rating of level 2 or higher on the Index of Treatment Refractory Depression
* Current diagnosis of any of the following psychiatric disorders: psychotic or organic mental, bipolar, primary obsessive compulsive, borderline personality, antisocial personality, or eating
* Current diagnosis of comorbid chronic depression that is disabling
* Current substance abuse
* Score less than 14 on the Hamilton Rating Scale for Depression-17 (HRSD-17)
* At risk for suicide
* Pregnancy or plan to become pregnant during the study
* Practice meditation more than once a week or yoga more than twice a week at study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2004-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Relapse of depression | Measured at Month 18

CONTACTS AND LOCATIONS:
Overall Officials: Zindel V. Segal, PhD, Principal Investigator — Center for Addiction and Mental Health
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

REFERENCES:
- [Background] Teasdale JD, Segal ZV, Williams JM, Ridgeway VA, Soulsby JM, Lau MA. Prevention of relapse/recurrence in major depression by mindfulness-based cognitive therapy. J Consult Clin Psychol. 2000 Aug;68(4):615-23. doi: 10.1037//0022-006x.68.4.615. PMID 10965637
- [Background] Ma SH, Teasdale JD. Mindfulness-based cognitive therapy for depression: replication and exploration of differential relapse prevention effects. J Consult Clin Psychol. 2004 Feb;72(1):31-40. doi: 10.1037/0022-006X.72.1.31. PMID 14756612
- [Background] Teasdale JD, Moore RG, Hayhurst H, Pope M, Williams S, Segal ZV. Metacognitive awareness and prevention of relapse in depression: empirical evidence. J Consult Clin Psychol. 2002 Apr;70(2):275-87. doi: 10.1037//0022-006x.70.2.275. PMID 11952186
- [Background] Segal ZV, Pearson JL, Thase ME. Challenges in preventing relapse in major depression. Report of a National Institute of Mental Health Workshop on state of the science of relapse prevention in major depression. J Affect Disord. 2003 Nov;77(2):97-108. doi: 10.1016/s0165-0327(02)00112-x. PMID 14607387
- [Background] Segal ZV, Bieling P, Young T, MacQueen G, Cooke R, Martin L, Bloch R, Levitan RD. Antidepressant monotherapy vs sequential pharmacotherapy and mindfulness-based cognitive therapy, or placebo, for relapse prophylaxis in recurrent depression. Arch Gen Psychiatry. 2010 Dec;67(12):1256-64. doi: 10.1001/archgenpsychiatry.2010.168. PMID 21135325
- [Background] Bieling PJ, Hawley LL, Bloch RT, Corcoran KM, Levitan RD, Young LT, Macqueen GM, Segal ZV. Treatment-specific changes in decentering following mindfulness-based cognitive therapy versus antidepressant medication or placebo for prevention of depressive relapse. J Consult Clin Psychol. 2012 Jun;80(3):365-72. doi: 10.1037/a0027483. Epub 2012 Mar 12. PMID 22409641